CLINICAL TRIAL: NCT01649063
Title: Principle Investigator
Brief Title: Comparing the Shape and Frequency of Uterine Contractions
Status: Completed | Type: Observational
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Samira Ebrahimzadeh Zagami, School of Nursing & Midwifery, Mashhad University of Medical Sciences
Other Study IDs: vaginal delivery and cesarean
Record Dates: First submitted 2012-07-21; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Uterine Contractions; Delivery
Keywords: Uterine contraction;; Shape; Frequency;; First stage labor;; Fall; Rise ratio.

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- the shape and frequency of uterine contractions in delivery: Uterine contractions were recorded by using fetal monitoring system (Model FC1400) at the beginning of the active phase (cervical dilatation 3-4 cm) for 30 min in two groups.
- the shape and frequency of uterine contractions in cesarean: Uterine contractions were recorded by using fetal monitoring system (Model FC1400) at the beginning of the active phase (cervical dilatation 3-4 cm) for 30 min in two groups.

SUMMARY:
Dystocia is the most common indication for primary cesarean section. The most common cause of dystocia is uterine dysfunction. In all cephalopelvic disproportion studies, more attention is usually paid on fetus and pelvic rather than on the role of uterine contraction in delivery. So we decided to determine the relationship between dystocia and uterine contraction patterns.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 years
* singleton pregnancy with cephalic term presentation
* tendency to do vaginal delivery
* having no medical or mental diseases
* having no pregnancy complications
* Intact membranes
* BMI<26

Exclusion Criteria:

* using oxytocin before and during the monitoring of contractions
* performing cesarean section for any reason except arrested delivery or pelvic constriction
* the birth weight< 2500 or >4000
* using the analgesia such as epidural anesthesia morphine and pethidine during the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primiparous women
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
the shape and frequency of uterine contractions | up to 15 months
  Uterus contractions were recorded using electronic fetal monitoring at the beginning of the active phase of labor (dilatation 3-5 cm) for 30 min.